CLINICAL TRIAL: NCT03477019
Title: Ultrasound-enhanced Delivery of Chemotherapy to Patients With Liver Metastasis From Breast- and Colorectal Carcinoma- a Randomized Trial
Brief Title: Ultrasound-enhanced Delivery of Chemotherapy to Patients With Liver Metastasis From Breast- and Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/13; 2018-002814-11 (EudraCT Number)
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Neoplasms; Breast Neoplasms
Keywords: Contrast Agent BR; SonoVue; Ultrasonic Therapy; Neoplasm Metastasis; Liver; Microbubbles
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — contrast agent BR1

STUDY DESIGN:
Intervention Model Description: Two liver metastases in every patient are preselected on baseline computer tomography. These will be randomized to either 1) target lesion to be treated or 2) control lesion. Difference in response (pre- and post-treatment measure) between treated lesions and control lesions will be the primary outcome of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breast cancer target lesion (Experimental): This arm will receive experimental treatment of focused ultrasound. In addition this arm will receive treatment with microbubbles intravenously and conventional chemotherapy for breast cancer.
  Interventions: Drug: SonoVue; Procedure: Focused Ultrasound
- Breast cancer control lesion (Other): This arm will only receive treatment with conventional chemotherapy for breastcancer and microbubbles intravenously.
  Interventions: Drug: SonoVue
- Colorectal cancer target lesion (Experimental): This arm will receive experimental treatment of focused ultrasound. In addition this arm will receive treatment with microbubbles intravenously and conventional chemotherapy for colorectal cancer.
  Interventions: Drug: SonoVue; Procedure: Focused Ultrasound
- Colorectal cancer control lesion (Other): This arm will only receive treatment with conventional chemotherapy for colorectal cancer and microbubbles intravenously.
  Interventions: Drug: SonoVue

INTERVENTIONS:
Drug: SonoVue — consists of microbubbles containing sulfur hexafluoride stabilized by phospholipids.
  Bolus doses à 1,0ml administered every 3.5 minutes , repeated 9 times. Total duration of treatment: 31,5 minutes. This treatment will be repeated maximally 4 times at 2 or 3 week intervals, depending on the patient's diagonse and treatment protocol.
Procedure: Focused Ultrasound — ultrasound pulses will be generated by a clinically approved ultrasound skanner and probe.
  Arms: Breast cancer target lesion; Colorectal cancer target lesion

SUMMARY:
The aim of this clinical trial is to investigate whether the therapeutic response of chemotherapy can be improved by focused ultrasound and microbubbles. Patients with liver metastases from breast cancer and colorectal cancer will be included. Computer Tomography (CT) will be performed as a baseline scan before treatment start. Two metastases in each patients liver will be preselected and randomized to either "target lesion" to be treated or "control lesion" to serve as internal control. The patients will receive conventional treatment with chemotherapy according to national guidelines. After intravenous chemotherapy infusion the patients will receive the experimental treatment. The target lesion will get focused ultrasound (FUS). Simultaneously repeated bolus-doses of microbubbles will be administered intravenously. The investigators will measure the difference in response between FUS- treated and -untreated lesions on the post-treatment CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified breast carcinoma or colorectal carcinoma
* 2 or multiple liver metastases
* considered eligible by a consulting oncologist for first line treatment with chemotherapy in the group of taxanes (patients with breast cancer) or the combination regimen FOLFIRI (patients with colorectal carcinoma)
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations

Exclusion Criteria:

* Known contraindications for ultrasound contrast-enhancement agent Sonovue® (Bracco)
* Hematological bleeding status before experimental treatment: Hb < 8g/dL, trc < 80 x109/l, APTT˃ 45s, INR ˃ 1,5
* Considered eligible for surgical removal of liver metastases
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
difference in measured response between treated and untreated lesions | From baseline examination CT to response evaluation CT: 10-12 weeks
  Response is measured in change in size of the treated metastases.

SECONDARY OUTCOMES:
Occurrence of adverse effects | 8 weeks
  questionnaire 'Common toxicity criteria'

CONTACTS AND LOCATIONS:
Overall Officials: Arne Solberg, PhD, MD, Study Director — St. Olavs Hospital
Locations (1):
- St.Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Yes.Individual participant data that underlie the results reported in this article, after deidentification(text, tables, figures, and appendices). Protocol can be shared beginning 3 months and ending 5 years following article publication. Interested researchers who provide a reasonable, sound proposal are encouraged to direct this to the first author.